CLINICAL TRIAL: NCT04488380
Title: Clinical Performance of Glass Ionomer Versus Resin Composite Restorations Performed Without Rubber-Dam Isolation
Brief Title: Clinical Performance of Glass Ionomer Versus Resin Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Huseyin Hatirli, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Restorative Glass Ionomer
Record Dates: First submitted 2020-07-13; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Dental Caries
Keywords: restorative glass ionomer
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: One of the Glass ionomer restorative or Resin composite restorative materials were applied to carious mandibular 2nd molar teeth.
Who Masked: Outcomes Assessor

ARMS (2):
- high-viscosity glass ionomer restoration (Experimental): One of the carious mandibular 2nd molar teeth (according to randomisation) will be restored with high-viscosity glass ionomer restoration (Equia, GC)
  Interventions: Other: dental restoration
- nano-hybrid composite resin (Experimental): One of the carious mandibular 2nd molar teeth will be restored with nano-hybrid composite resin (GrandioSO, Voco)
  Interventions: Other: dental restoration

INTERVENTIONS:
Other: dental restoration — Restoration of carious mandibular 2nd molar teeth either with high viscosity glass ionomer or nanohybrid composite resin

SUMMARY:
The aim of this randomised-controlled, single-blind, split-mouth, and single-centre clinical trial was to evaluate the 2-year clinical performances of a high-viscosity glass ionomer and nanohybrid composite resin in occlusal restorations on mandibular second molar teeth in patients at risk for salivary contamination.

DETAILED DESCRIPTION:
Occlusal carious lesions on the right and left mandibular second molars of 56 patients (26 females, 30 males) were restored in a split-mouth design. A high-viscosity glass ionomer (Hv-GIC) (Equia, GC) was used to restore the carious lesions in patients in the treatment group, while a nano-hybrid composite resin (GSO) (GrandioSO, Voco) was used for patients in the control group. Clinical evaluations of the restorations were performed at 1-week, 6-month, 1-year, and 2-year follow-up appointments, according to the FDI criteria. Data were analysed using the Friedman's analysis of variance and Mann-Whitney U tests (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

* good health and oral hygiene,
* occlusal carious lesions on both mandibular second molars,
* mandibular second molars with mesial and occlusal contacts,
* contraindication to the use of rubber dam,
* the ability to return for periodic follow-up visits.

Exclusion Criteria:

* restoration on mandibular second molars.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Surface lustre of dental restorations | Changes of dental restorations regarding surface lustre were observed at 1-week, 6-month, 1-year, and 2-year results were compared between two restorative material and change of material suring the study is observed
  Surface lustre of dental restorations were observed by visual examination of two examiners. Restorations were scored 1 to 5 according to FDI criteria (1. Lustre comparable to enamel, 2. Slightly dull, not noticeable from speaking distance, 3.Dull surface but acceptable if covered with film of saliva, 4. Rough surface, cannot be masked by saliva film, simple polishing is not sufficient. Further intervention necessary, 5. Very rough, unacceptable plaque retentive surface.).
Staining restoration surface and restoration margin | Changes of dental restorations regarding surface lustre were observed at 1-week, 6-month, 1-year, and 2-year results were compared between two restorative material and change of material suring the study is observed
  Surface lustre of dental restorations were observed by visual examination of two examiners. Restorations were scored 1 to 5 according to FDI criteria (1. No surface staining, no marginal staining, 2. Minor surface staining, minor marginal staining easily removable by polishing, 3. oderate surface staining and moderate marginal staining that may also present on other teeth, not esthetically unacceptable, 4. Unacceptable surface staining on the restoration and major intervention necessary for improvement and Pronounced marginal staining; major intervention necessary for improvement, 5. Severe surface staining and/or subsurface staining, generalized or localized, not accessible for intervention and deep marginal staining, not accessible for intervention.).
Fracture of material and retention | Changes of dental restorations regarding Fracture of material and retention were observed at 1-week, 6-month, 1-year, and 2-year results were compared between two restorative material and change of material suring the study is observed
  Fracture of material and retention of dental restorations were observed by visual examination of two examiners. Restorations were scored 1 to 5 according to FDI criteria (1. No fractures / cracks, 2. Small hairline crack. 3. Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact, 4. Material chip fractures which damage marginal quality or, approximal contacts. 5. (Partial or complete) loss of restoration or multiple fractures.).
Recurrence of caries | Changes of dental restorations regarding recurrence of caries were observed at 1-week, 6-month, 1-year, and 2-year results were compared between two restorative material and change of material suring the study is observed
  Recurrence of caries were observed by visual examination of two examiners. Restorations were scored 1 to 5 according to FDI criteria (1. No secondary or primary caries 2. Small and localized. 3 Larger areas of 1. Demineralisation 2. Erosion or 3. Abrasion/abfraction, dentine not exposed Only preventive measures necessary 4. Caries with cavitation and suspected undermining caries Localized and accessible can be repaired, 5. Deep caries or exposed dentine that is not accessible for repair of restoration.)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gurgan S, Kutuk ZB, Yalcin Cakir F, Ergin E. A randomized controlled 10 years follow up of a glass ionomer restorative material in class I and class II cavities. J Dent. 2020 Mar;94:103175. doi: 10.1016/j.jdent.2019.07.013. Epub 2019 Jul 25. PMID 31351909
- [Background] Turkun LS, Kanik O. A Prospective Six-Year Clinical Study Evaluating Reinforced Glass Ionomer Cements with Resin Coating on Posterior Teeth: Quo Vadis? Oper Dent. 2016 Nov/Dec;41(6):587-598. doi: 10.2341/15-331-C. Epub 2016 Aug 29. PMID 27571238
- [Derived] Hatirli H, Yasa B, Celik EU. Clinical performance of high-viscosity glass ionomer and resin composite on minimally invasive occlusal restorations performed without rubber-dam isolation: a two-year randomised split-mouth study. Clin Oral Investig. 2021 Sep;25(9):5493-5503. doi: 10.1007/s00784-021-03857-0. Epub 2021 Mar 8. PMID 33683465